CLINICAL TRIAL: NCT01073280
Title: Cerebral, Meningeal Biopsy by Flexible Endoscopy in Patients Without Neurological Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Responsible Party: Cerebral , meningeal biopsy by flexibel endoscopy in patients without neurological diagnosis, UASLP
Other Study IDs: NCT150210
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2010-02

CONDITIONS: Neurological Disease
Keywords: Cerebral and subarachnoid biopsy; flexible endoscopy; Patients with neurological findings without diagnosis.
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- undeterminated neurological disease, cerebral endoscopy: patients without neurological diagnosis that require cerebral , meningeal diagnosis
  Interventions: Procedure: cerebral flexible endoscopy

INTERVENTIONS:
Procedure: cerebral flexible endoscopy — The investigators will make a burrhole in the precoronal suture introducing the flexible endoscope taking a cerebral and a basal meningeal biopsy

SUMMARY:
The investigators will take cerebral and subarachnoid biopsy by flexible endoscopy in patients without neurological findings. The investigators will use retrospective and prospective patients.

DETAILED DESCRIPTION:
Test the useful of the flexible endoscopy in patients without neurological diagnosis.

Developed a diagnosis method for idiopathic neurological findings.

Compare the cerebral and subarachnoid biopsy each other

ELIGIBILITY:
Inclusion Criteria:

* patients with neurological disease and with out diagnosis

Exclusion Criteria:

* death of the patient
* patients with neurological diagnosis

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients between 0 and 85years old with neurological diseases that there are not a diagnosis
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-01 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Test the useful of the cerebral and subarachnoid biopsy by flexible endoscopy in patients without neurological findings | 2 weeks

SECONDARY OUTCOMES:
Developed a diagnosis method for idiopathic neurological findings. Compare the cerebral and subarachnoid biopsy each other | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Central Dr. Ignacio Morones Prieto, San Luis Potosí City, San Luis Potosí, Mexico